CLINICAL TRIAL: NCT04764773
Title: Persistence of Symptoms After Improvement of Acute COVID19 Infection in Sohag Governorate, Egypt, A Longitudinal Study
Brief Title: Persistence of Symptoms After Improvement of Acute COVID-19
Acronym: COVID-19
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mona Mohammed Abdelrhman, Principal investigator, Sohag University
Other Study IDs: Soh-Med-21-02-46
Record Dates: First submitted 2021-02-19; First posted 2021-02-21 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-11

CONDITIONS: Corona Virus Infection
Keywords: Persistent symptoms; Recovery; COVID-19
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: Patient who had COVID19 infection
  Interventions: Other: No intervention
- control: healthy volunteer who were age and sex matched with our patients
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Coronavirus disease pandemic has been started in late 2019. Survivors of COVID-19 are significantly more likely to develop clinical sequelae three months after discharge from the hospital than those without COVID-19 infection. This is true not only for general and respiratory symptoms but also for cardiovascular and psychosocial symptoms. This suggests that these symptoms may indeed be the sequelae of recovery for COVID-19 survivors. So, we aimed to detect the prevalence and to evaluate the type of symptoms that could persist after the recovery from COVID19 infection in Sohag governorate, Egypt.

DETAILED DESCRIPTION:
About one hundred patients who were test positive for SARS-CoV2 and were improved and discharged from Sohag isolation hospitals and isolation department for COVID19 in Sohag University hospitals during the period from 15th May, 2020 to 25th July, 2020 will be included in our study. Patient improvement and discharge criteria include 10 day from symptoms onset in addition to 3 day free of fever and respiratory symptoms.

Patients with severe complex illness, pregnant or lactating females and patient who refuse to participate or give complete detailed history will be excluded from the study.

The study protocol will be approved by the scientific Research Ethical committee, Faculty of Medicine, Sohag University A control group of healthy volunteer who were age and sex matched to our patient were included

After taken informed consent according to Sohag University Ethical Committee, the baseline data will be collected from Sohag isolation hospital of COVID19, then the researchers will perform interviews with all participants through mobile phone. The interview will include:

* Name (Optional)
* Age
* Sex
* Occupation
* Presence of DM, HTN or any chronic illness
* Asking about Smoking
* The date of catching COVID19 infection
* Asking about symptoms of COVID19 infection and duration of each symptom.
* Asking about any residual symptoms as: Fatigue, Myalgia, Arthralgia, Chest pain, Dyspnea, Dry cough, Productive cough, Sore Throat, Anosmia, Loss of taste sensation, Nausea, Anorexia, Diarrhea, Redness of the eye, Headache, Confusion and Depression

Statistical analysis:

Data will be analyzed using STATA version 14.2 (Statistical Software: Release 14.2 College Station, TX: Stata Corp LP). Quantitative data will be represented as mean, standard deviation, median and range. normally distributed. Qualitative data will be presented as numbers and percentages. Chi square test will be used for comparison of percentages in different groups. P value will be considered significant if it was less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

Positive for SARS-CoV2

Exclusion Criteria:

* Patients with severe complex illness, pregnant or lactating females and patient who refuse to participate or give complete detailed history

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients who were test positive for SARS-CoV2 and were improved and discharged from Sohag isolation hospitals and isolation department for COVID19 in Sohag University hospitals
Sampling Method: Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Percentage of patient who had persistent symptoms after recovery of acute covid19 | during the period from 15th May,2020 to the end of February, 2021
Type of persistent symptom after acute covid19 | during the period from the start of June 2020 to the end of July 2020
Risk factors for persistent symptoms after recovery of acute covid19 | during the period from 15th May,2020 to the end of February, 2021

CONTACTS AND LOCATIONS:
Overall Officials: Noha Abdelrahman, assistant-lecturer, Study Chair — Sohag University
Locations (1):
- Mona Mohammed Abdelrahman, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xiong Q, Xu M, Li J, Liu Y, Zhang J, Xu Y, Dong W. Clinical sequelae of COVID-19 survivors in Wuhan, China: a single-centre longitudinal study. Clin Microbiol Infect. 2021 Jan;27(1):89-95. doi: 10.1016/j.cmi.2020.09.023. Epub 2020 Sep 23. PMID 32979574
- [Derived] Abdelrahman MM, Abd-Elrahman NM, Bakheet TM. Persistence of symptoms after improvement of acute COVID19 infection, a longitudinal study. J Med Virol. 2021 Oct;93(10):5942-5946. doi: 10.1002/jmv.27156. Epub 2021 Jul 2. PMID 34171139